CLINICAL TRIAL: NCT03237936
Title: A Phase IV, Prospective, Open-label, Multicentre, Single Arm, 3-month Proof of Concept Study to Assess the Effect of IKERVIS® Eye Drops Administered Once Daily on the Quality of Vision in Dry Eye Disease (DED) Patients With Severe Keratitis
Brief Title: Effect of IKERVIS® Eye Drops Once Daily on the Quality of Vision in Dry Eye Disease Patients With Severe Keratitis
Acronym: FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVG16E128
Record Dates: First submitted 2017-01-13; First posted 2017-08-03 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Keratitis
MeSH Terms: conditions — Keratitis | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IKERVIS® (1mg/mL ciclosporin) eye drops (Experimental): one drop of study medication (IKERVIS®1mg/mL) once daily in each eye at bedtime during 3 months.
  Interventions: Drug: 1mg/mL ciclosporin

INTERVENTIONS:
Drug: 1mg/mL ciclosporin — IKERVIS® (1mg/ml ciclosporin) eye drops administered once daily following 3 months of treatment
  Other Names: IKERVIS®

SUMMARY:
The proposed 3-month study is a prospective, open-label, multicentre, phase IV, proof of concept study. The study is designed to assess the effect on the quality of vision of IKERVIS® (1mg/mL ciclosporin) eye drops administered once daily in dry eye disease (DED) patients with severe keratitis, as well as its safety and efficacy.

DETAILED DESCRIPTION:
In this phase IV clinical trial the Month 3 visit assessments will be used to assess the efficacy (quality of vision and other parameters) and safety of IKERVIS® in DED patients with severe keratitis.

To assess the effect on the quality of vision of IKERVIS® (1mg/ml ciclosporin) eye drops administered once daily in adult dry eye disease (DED) patients with severe keratitis over 3 months of treatment.

To assess the safety of DED patients with severe keratitis treated with IKERVIS® (1mg/mL ciclosporin) for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility is determined according to the following criteria:

  1. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements.
  2. The patient signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures
  3. Male or female patient is aged 18 years or above.
  4. DED patients with persistent severe keratitis at the Screening and

     Baseline Visits defined as the following:

     • CFS score of 3, 4 or 5 on the modified Oxford scale
  5. Patient must be willing and able to undergo and return for scheduled study-related examinations.
  6. The same eye (eligible eye) should fulfill all the above criteria.

Exclusion Criteria:

* Patients with history of ocular trauma or ocular infection (viral, bacterial, fungal, protozoal) within 90 days before the Screening Visit and any ocular diseases other than dry eye disease requiring topical ocular treatment during the course of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean PISELLA, Principal Investigator — CHU Bretonneau
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IKERVIS® (1mg/mL Ciclosporin) Eye Drops
Started | 17
Completed | 16
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | IKERVIS® (1mg/mL Ciclosporin) Eye Drops
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 17

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between the Change From Baseline in VMR Measured With FVA System at Month 3 and the Change From Baseline in the CFS at Month 3.
Description: Spearman's coefficient of correlation will be calculated at Month 3 between the change from baseline of Corneal Fluorescein Staining (CFS) and respectively the change from baseline of Visual Maintenance Ratio (VRM).
Time Frame: at month 3
Measure: Number (95% Confidence Interval); unit: Spearman's coefficient of correlation
Arm/Group | IKERVIS® (1mg/mL Ciclosporin) Eye Drops
Number analyzed (Participants) | 17
Spearman's coefficient of correlation | -0.7028 [-0.8797 to -0.3158]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until the subject's participation in the study ended at Month 3.
Description: Adverse events (AEs) are presented for the Safety analysis population. AEs were defined as any untoward medical occurrence in the study irrespective of a causal relationship with the study medication.
Arm/Group | IKERVIS® (1mg/mL Ciclosporin) Eye Drops
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IKERVIS® (1mg/mL Ciclosporin) Eye Drops (N=17)
EYE IRRITATION (Eye disorders) | 3
DRY EYE (Eye disorders) | 2
EYE BURNS (Eye disorders) | 1
EYELID OEDEMA (Eye disorders) | 1
PHOTOPHOBIA (Eye disorders) | 1
VISUAL ACUITY REDUCED (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03237936/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03237936/SAP_001.pdf